CLINICAL TRIAL: NCT03135054
Title: A Phase II Single-arm Open-labeled Study Evaluating Combination of Quizartinib and Omacetaxine Mepesuccinate (QUIZOM) in Newly Diagnosed or Relapsed/Refractory AML Carrying FLT3-ITD
Brief Title: Combination of Quizartinib and Omacetaxine Mepesuccinate for AML Carrying FLT3-ITD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Anskar Y.H. Leung, Clinical Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AML005
Record Dates: First submitted 2017-04-26; First posted 2017-05-01 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: AML; FLT3-ITD Mutation
Keywords: FLT3-ITD (+) AML; Quizartinib, Omacetaxine mepesuccinate
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — quizartinib; Homoharringtonine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination (Experimental): Quizartinib is a second generation FLT3 inhibitors.The starting dose of quizartinib will be 30 mg/day oral unless the patients are taking a strong CYP3A4 inhibitor in which case the dose will be 20 mg /day. Quizartinib should be taken continuously throughout the treatment period unless there is no evidence of response at first assessment on day 28 or progressive disease at any time during the treatment.
  Omacetaxine Mepesuccinate will be given at 1.5 mg/m2/day (maximum dose 3 mg) for 7 days (concurrently with quizartinib) in 28-day cycle.
  Interventions: Drug: Quizartinib; Drug: Omacetaxine Mepesuccinate Injection

INTERVENTIONS:
Drug: Quizartinib — Quizartinib is an oral FLT3 receptor tyrosine kinase inhibitor
  Other Names: AC220
Drug: Omacetaxine Mepesuccinate Injection — Omacetaxine Mepesuccinate is a pharmaceutical drug substance that is indicated for treatment of chronic myeloid leukemia (CML)
  Other Names: homoharringtonine

SUMMARY:
The study aims to test if combination of quizartinib (AC220) and omacetaxine mepesuccinate (OM, also known as homoharringtonine) results in durable composite complete remission (CRc) in patients with newly diagnosed or relapsed/refractory (R/R) acute myeloid leukemia (AML) carrying FLT3-ITD (Fms-Like Tyrosine Kinase 3 - Internal Tandem Duplication).

DETAILED DESCRIPTION:
The type of AML being studied in this clinical trial is known as FMS-like tyrosine kinase 3 (FLT3)-internal tandem duplication (ITD) positive AML. This type of AML has an alteration (or mutation) in genes, which may associated with high risk of relapse after conventional chemotherapy and hence an extremely poor clinical outcome.

Second generation FLT3 inhibitors including quizartinib are effective in inducing remission. However, their effects are only transient. There is an unmet clinic need to enhance their effectiveness, hence clinical application.

This is a Phase II single-arm open-labeled study. A total of 40 eligible patients with consent will be recruited, including 20 patients with newly diagnosed and 20 with R/R FLT3-ITD AML. For newly diagnosed patients, diagnostic bone marrow (BM) and/or peripheral blood (PB) will be evaluated by next generation sequencing (NGS) based on myeloid panel that comprises 54 myeloid genes as well as their in vitro response to QUIZOM based on an in-house platform that was established in our laboratory. FLT3-ITD allelic burden will also be evaluated. For R/R patients, FLT3-ITD status and allelic burden will be confirmed before QUIZOM treatment. Both groups of patients will receive quizartinib 30 mg daily continuously and OM 1.5 mg/m2 daily for 7 days every 28 days until progression or allogeneic hematopoietic stem cell transplantation (HSCT). BM examination will be performed on day 21 to document morphological response and FLT3-ITD allelic burden. At leukemia progression, BM and/or PB samples will be collected and their in vitro response to QUIZOM examined. The tyrosine kinase domain (TKD) of FLT3 will also be sequenced and FLT3-ITD allelic burden will be evaluated.

Eligible patients will receive QUIZOM comprising quizartinib and OM. The starting dose of quizartinib will be 30 mg/day unless the patients are taking a strong CYP3A4 inhibitor in which case the dose will be 20 mg /day. Quizartinib should be taken continuously throughout the treatment period unless there is no evidence of response at first assessment on day 21 or progressive disease at any time during the treatment.

OM will be given at 1.5 mg/m2/day (maximum dose 3 mg) for 7 days (concurrently with quizartinib) in 28-day cycle. QUIZOM will be continued until leukemia progression or allogeneic HSCT. Thereafter, patients will be followed up and information about disease status and survival will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent approved by the Institutional Review Board (IRB).
2. Age ≥18 years
3. Documented primary AML or AML secondary to myelodysplastic syndrome (MDS), as defined by World Health Organization criteria
4. At diagnosis or in morphological relapse after an initial remission or refractory after induction chemotherapy, with or without HSCT
5. Documentation of FLT3-ITD in BM or blood with allelic burden of ≥ 20% as determined by the study site laboratory
6. ECOG performance score 0-2
7. Discontinuation of prior AML treatment ≥ 2 weeks before the start of QUIZOM (except hydroxyurea or other treatment to control leukocytosis).
8. Serum creatinine ≤1.5×upper limit of normal (ULN), or glomerular filtration rate >25 mL/min, as calculated with the Cockcroft-Gault formula.
9. Serum potassium, magnesium, and calcium (corrected for albumin) within institutional normal limits. Subjects with electrolytes outside the normal range will be eligible if these values are corrected upon retesting following any necessary supplementation.
10. Total serum bilirubin ≤1.5×ULN.
11. Serum aspartate transaminase (AST) and/or alanine transaminase (ALT) ≤ 2.5×ULN.

Exclusion Criteria:

1. Acute promyelocytic leukemia (AML subtype M3)
2. Prior treatment with any FLT3 inhibitors
3. Known infection with human immunodeficiency virus, or active hepatitis B or C infection.
4. Refusal of blood product transfusion.
5. Uncontrolled or significant cardiovascular disease, including:

   i. QTcF interval > 450 msec ii. Bradycardia of ≤ 50 BPM iii. Diagnosed or suspected long QT syndrome, or known family history of long QT syndrome iv. History of clinically relevant ventricular arrhythmias, such as ventricular tachycardia, ventricular fibrillation, or torsade de pointes v. History of second or third degree heart block. Candidates with a history of heart block may be eligible if they currently have pacemakers, and have no history of fainting or clinically relevant arrhythmia with pacemakers.

   vi. Myocardial infarction within 6 months prior to screening vii. Uncontrolled angina pectoris within 6 months prior to screening viii. New York Heart Association (NYHA) Class 3 or 4 congestive heart failure ix. Uncontrolled hypertension x. Complete left or right bundle branch block
6. In a man whose sexual partner is a woman of childbearing potential, unwillingness or inability of the man or woman to use an acceptable contraceptive method for the entire study treatment period and for at least 3 months after study treatment completion
7. In a heterosexually active woman of childbearing potential, unwillingness or inability to use an acceptable contraceptive method for the entire study treatment period and for at least 3 months after study treatment completion
8. Pregnancy
9. Female subjects must agree not to breastfeed at screening and throughout the study period, and for 45 days after the final study drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Complete remission | up to 16 weeks
  No increase in blasts in BM or PB (<5% of total nucleated cells), with absolute neutrophil count ≥ 1x109/L and platelet count ≥ 100 x109/L

CONTACTS AND LOCATIONS:
Overall Officials: Anskar Leung, Professor, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided